# **Protocol Title**

# Respiratory virus infections in acutely hospitalized adult patients with pulmonary and extrapulmonary complications

# **Principal Investigator**

Dr. Kelvin To MBBS, FRCPath, FHKCPath, FRCP (Edin), MD

> Date: 4<sup>th</sup> January 2019 Version: 20190104

# **Table of content**

| Section | Content | Page number |
|---|---|---|
| 1 | Protocol synopsis | 3 |
| 2 | Background and rationale | 4 |
| 2.1 | Background of respiratory virus infection | 4 |
| 2.2 | Study rationale | 4 |
| 3 | Study Design | 5 |
| 3.1 | Study objectives | 5 |
| 3.2 | Study design and organization | 5 |
| 3.2.1 | Overall study design | 5 |
| 3.3 | Outcome measurements | 6 |
| 3.3.1 | Primary outcome measurement | 6 |
| 3.3.2 | Secondary outcome measurements | 6 |
| 3.4 | Informed consent | 6 |
| 3.5 | Confidentiality of data | 6 |
| 3.6 | Archive of data | 7 |
| 4 | Selection and enrollment of participants | 7 |
| 4.1 | Selection of study population at in-patient | 7 |
| 4.11 | Inclusion criteria | 7 |
| 4.12 | Exclusion criteria | 7 |
| 4.2 | Selection of study population at out-patient | 7 |
| 4.2.1 | Inclusion criteria | 7 |
| 4.2.2 | Exclusion criteria | 7 |
| 4.3 | Study enrollment procedures | 8 |
| 5 | Study procedures | 8 |
| 5.1 | Schedule of evaluations | 8 |
| 5.1.1 | Participants at acute medical ward (inpatients) | 8 |
| 5.1.2 | Participants at the out-patient clinic | 8 |
| 5.2 | Assessment and clinical data collection | 8 |
| 5.3 | Detection of respiratory viruses | 9 |
| 5.3.1 | Specimen collection | 9 |
| 5.3.2 | Molecular testing of respiratory viruses | 9 |
| 5.4 | Healthcare utilization of respiratory virus infection | 9 |
| 6 | Statistical methods | 10 |
| 6.1 | Sample size | 10 |
| 6.2 | Analysis of study | 10 |
| 7 | Study team and study site | 11 |
| 7.1 | Study team | 11 |
| 7.2 | Study site | 11 |
| 8 | References | 11 |

# 1. PROTOCOL SYNOPSIS:

| Protocol title | Respiratory virus infections in acutely hospitalized adult patients with pulmonary and extrapulmonary complications |
|---|---|
| Hypothesis | The incidence of respiratory virus infection were underestimated |
| Primary objective | To determine the incidence and adjusted population attributable fraction of respiratory virus infection among patients with pulmonary and extrapulmonary complications |
| Study participants | Adult hospitalized patients admitted to the acute medical ward of Queen Mary Hospital Adult out-patients of Queen Mary Hospital |
| Study design | This is a prospective cohort study involving hospitalized adult patients admitted to the acute medical ward of Queen Mary Hospital, an acute care university-affiliated hospital with 1,700 beds in Hong Kong. Consecutive patients will be screened for eligibility based on inclusion and exclusion criteria. Written informed consent will be obtained from all study participants. Saliva specimens will be collected from study participants, and will be tested for respiratory viruses by a multiplex PCR panel. Patients' demographics, underlying diseases, and outcome measures will be collected. The crude incidence will be assessed. Adjusted population attributable fraction will be calculated by adjusting the crude incidence of acutely hospitalized adult patients with the background rate among adult out-patients. |
| Primary outcome | Incidence of respiratory viruses |
| Secondary outcome | <ol> <li>Length of hospital stay</li> <li>Length of stay in general medical ward</li> <li>Length of stay in high dependency unit</li> <li>Length of stay in intensive care unit</li> <li>Proportion of patients requiring oxygen supplementation</li> <li>Proportion of patients requiring positive pressure ventilation</li> <li>Proportion of patients requiring intubation</li> <li>Proportion of patients admitted to intensive care unit</li> <li>Proportion of patients admitted to coronary care unit</li> <li>Proportion of patients admitted to high dependency unit</li> <li>Proportion of patients who die during hospitalization</li> <li>Initial blood test results on admission</li> <li>Radiological investigation results</li> <li>Microbiological investigations results</li> </ol> |
| Data analysis | The fraction of hospitalization that can be attributed by a particular respiratory pathogen will be calculated using adjusted population attributable fraction. |

Continuous variables and categorical variables will be compared using Mann Whitney U test and Fisher's exact test, respectively. A *P* value of <0.05 with two sided testing will be considered statistically significant. Statistical test will be performed using SPSS 23.0.0.

#### 2. BACKGROUND AND RATIONALE

# 2.1. Background and study rationale

Respiratory viruses cause severe infections, and contribute to a substantial number of hospitalizations, admission to intensive care units and deaths (1). Many hospitalizations due to respiratory virus infection are related to pneumonia or exacerbation of chronic lung disease. In addition, many hospitalizations are related to extrapulmonary complications, such as acute coronary syndrome or stroke (2).

Previous studies have reported the incidence of respiratory viruses among patients with pulmonary complications (3), or the association of respiratory viruses with acute coronary syndrome or stroke (4). However, there are several problems associated with these studies. First, many of these studies are retrospective in nature, and therefore testing was only performed in selected patients with respiratory symptoms. Hence, many patients without respiratory symptoms were not recruited. Second, respiratory virus can be detected in some asymptomatic individuals. Therefore, the presence of respiratory virus may be an incidental finding rather than the cause of the complication. Third, many studies only focus on a few respiratory viruses, especially on influenza virus.

This study aims to address these issues. We propose to conduct a prospective cohort study. We will recruit hospitalized adult patients with exacerbation of underlying lung disease, acute coronary syndrome or stroke. As controls, we will recruit outpatients follow-up for chronic heart disease, chronic lung disease or neurological conditions. We will collect saliva from study participants and perform respiratory virus testing using a multiplex PCR panel. Our previous studies have shown that there is a high concordance between results from respiratory virus testing on saliva and nasopharyngeal specimens (5, 6).

Our study will provide accurate data on the epidemiology of respiratory viruses in pulmonary and extrapulmonary complications. These data are important for clinicians, public health practitioners and scientists.

#### 3. STUDY DESIGN

#### 3.1. Study objectives

- 1. To determine the crude incidence of respiratory virus infection among patients with exacerbation of chronic lung disease, acute coronary syndrome or stroke
- 2. To determine the adjusted population attributable fraction of respiratory virus infection among patients with exacerbation of chronic lung disease, acute coronary syndrome or stroke

# 3.2 Study design and organization

# 3.2.1 Overall study design

This is a prospective cohort study involving hospitalized adult patients admitted to the acute medical ward of Queen Mary Hospital, an acute care university-affiliated hospital with 1,700 beds in Hong Kong. Patients will be screened for eligibility based on inclusion and exclusion criteria. Written informed consent will be obtained from all study participants. Saliva specimens will be collected from study participants, and will be tested for respiratory viruses using a multiplex PCR panel. Patients' demographics, underlying diseases, and outcome measures will be collected.

Since respiratory viruses can be detected in asymptomatic adults, we will also recruit outpatients followed up for a chronic condition to determine the frequency of respiratory viruses among these patients without any acute symptoms requiring hospitalization. We will adjust the crude incidence from this background rate.

# 3.3 Outcome measurements

## 3.3.1 Primary outcome measurement

1. Incidence of respiratory viruses

# 3.3.2 Secondary outcome measurements

- 1. Length of hospital stay
- 2. Length of stay in general medical ward
- 3. Length of stay in high dependency unit
- 4. Length of stay in intensive care unit
- 5. Proportion of patients requiring oxygen supplementation
- 6. Proportion of patients requiring positive pressure ventilation
- 7. Proportion of patients requiring intubation
- 8. Proportion of patients admitted to intensive care unit
- 9. Proportion of patients admitted to coronary care unit
- 10. Proportion of patients admitted to high dependency unit
- 11. Proportion of patients who die during hospitalization
- 12. Initial blood test results on admission
- 13. Radiological investigation results
- 14. Microbiological investigations results

# 3.4. Informed consent

The investigator or his/her representative will explain the nature of the study to the subjects, and answer all questions by the subjects regarding this study. Prior to any study-related screening procedures being performed on the subject, the informed consent statement will be reviewed and signed and dated by the subjects and the person who administered the informed consent.

#### 3.5 Confidentiality of data

Permission for direct access to a subject's data will be sought in writing by the investigator and from the subject as part of the informed consent procedure. This gives permission to examine, analyse, verify and reproduce any records and reports that are important to the evaluation of the study. Any party (e.g., domestic and foreign regulatory authorities, monitors and auditors) with direct access must take all reasonable precautions within the constraints of the applicable regulatory requirements to maintain the confidentiality of the subjects' identities and the Hospital Authority's proprietary

information. It is the monitor's responsibility to verify that each subject has consented, in writing, to direct access.

# 3.6 Archive of data

The investigator must retain all study documentation pertaining to the conduct of the study at the study site for a period of at least 5 years.

# 3.7 Ethical and administrative endorsement

The study was approved by the Institutional Review Board (IRB) of the University of Hong Kong and Hospital Authority (IRB reference number: to be added when approved)

#### 4. SELECTION AND ENROLLMENT OF PARTICIPANTS

# 4.1 Selection of study population at in-patient

#### 4.1.1. Inclusion criteria

- 1. Admitted to the acute medical ward of Queen Mary Hospital via the accident and emergency department
- 2. Aged 18 years or above
- 3. Hospitalized for less than 24 hours at the time of recruitment
- 4. Presented with exacerbation of underlying lung disease, acute coronary syndrome or stroke
- 5. Competent and agree to provide written informed consent

# 4.1.2 Exclusion criteria

- 1. Admitted to any hospitals in the past 14 days
- 2. Respiratory virus testing performed in the past 14 days
- 3. Antiviral against respiratory virus given within the past 14 days
- 4. Not sufficient saliva

# 4.2 Selection of study population at out-patient

#### 4.2.1 Inclusion criteria

- 1. Aged 18 years or above
- 2. Follow-up at out-patient clinic or at the physiotherapy department of Queen Mary Hospital
- 3. Competent and agree to provide written informed consent

#### 4.2.2 Exclusion criteria

- 1. Admitted to any hospitals in the past 14 days
- 2. Respiratory virus testing performed in the past 14 days
- 3. Antiviral against respiratory virus given within the past 14 days
- 4. Onset of new respiratory or non-respiratory symptoms within the past 14 days
- 5. Not sufficient saliva

# 4.3 Study enrollment procedures

Patients will be screened for eligibility by a research nurse. Reasons for ineligibility or non-participation of eligible candidates will be documented. A written informed consent will be signed by the patient.

#### 5. STUDY PROCEDURES

# 5.1 Schedule of evaluations

# 5.1.1 Participants at the acute medical ward (in-patients)

On the day of enrollment:

- Inclusion and exclusion criteria
- Written informed consent
- Demographic information
- Questionnaire on vaccine history and symptoms
- Collection of saliva specimen

Follow-up after patient discharge

- Hospitalization data (length of stay, laboratory and radiological tests, treatment)

# 5.1.2 Participants at the out-patient clinic

On the day of enrollment:

- Inclusion and exclusion criteria
- Written informed consent
- Demographic information
- Questionnaire on vaccine history and symptoms
- Collection of saliva specimen

# 5.2 Assessment and clinical data collection

Initial symptom assessment will be performed by trained research nurses at the medical or at outpatient clinics. At the time of enrollment, the following information will be collected from the patient by the research staff using a standard questionnaire:

- Symptoms and date of symptom onset
- Prior use of oseltamivir or zanamivir within 14 days
- Prior use of antibiotics within 14 days
- Attended out-patient clinic for the same illness
- Close contacts with respiratory symptoms in the past 7 days
- Receive influenza vaccine in the past season
- Receive pneumococcal vaccine

The following data will be extracted from the clinical management system:

- Age, sex, comorbidities
- National Early Warning Score (NEWS) at A&E (20) (respiration rate, oxygen saturation, need for supplemental oxygen, temperature, systolic blood pressure, heart rate, level of consciousness)
- Time of hospital admission and discharge
- Clinical findings
  - Underlying disease

- Clinical symptoms and signs during hospitalization
- Hematological, biochemical, microbiological, immunological, and radiological investigation results on admission
- Need for supplementary oxygen, positive pressure ventilation, intubation, admission to intensive care unit, coronary care unit or high dependency unit during the hospital stay
- Final diagnosis

# **5.3** Detection of respiratory viruses

# 5.3.1 Specimen collection

Patients will be asked to spit out saliva (~1 ml) into a sterile container and viral transport medium (VTM) will be added as we described previously (5, 6). The specimens will be transported to the laboratory and stored at -80°C until testing.

# 5.3.2 Molecular testing of respiratory virus

Saliva will be tested for respiratory viruses using a commercially available multiplex PCR panel.

#### 6. STATISTICAL METHODS

# 6.1. Sample size

The sample size is based on the feasibility of the budget. A total of 100 hospitalized patients and 100 out-patients will be recruited.

#### 6.2 Analysis of the study

Crude incidence of each respiratory virus and overall respiratory virus infection among hospitalized patients and out-patients will be estimated. To adjust for the background rate of respiratory virus detection among out-patients, we will calculate adjusted population attributable fraction (aPAF) as described previously (22). Conceptually, aPAF represents the fraction of hospitalization that can be attributed to a particular pathogen. Death rate of each detected respiratory virus and overall respiratory virus infection among patients in the acute medical wards will be estimated.

For symptomatology of respiratory viruses, frequencies and proportions of respiratory and non-respiratory symptoms for each respiratory virus and overall respiratory virus infection will be calculated.

Statistical test will be performed using SPSS version 23.0. A *P* value of <0.05 with two-sided testing will be considered statistically significant.

#### 7. STUDY TEAM and STUDY SITE

#### 7.1 Study team

Principal investigator

- Design of study, coordination and assessment of subjects for study enrollment, analysis of data, writing up

# Co-investigators

- Coordination and assessment of subjects for study enrollment Study nurse
- Subject enrollment, collection of clinical specimens, data collection

## 7.2 Study site

Queen Mary Hospital, Pokfulam Road, Pokfulam, Hong Kong Special Administrative Region, China

# 8. REFERENCES

- 1. **World Health Organization.** 2013. Research needs for the Battle against Respiratory Viruses (BRaVe). Available at http://www.who.int/influenza/patient\_care/clinical/BRaVe\_Research\_Agenda\_2013.pdf? ua=1. Accessed on November 20, 2017.
- 2. **Sellers SA, Hagan RS, Hayden FG, Fischer WA, 2nd.** 2017. The hidden burden of influenza: A review of the extra-pulmonary complications of influenza infection. Influenza Other Respir Viruses **11:**372-393.
- 3. To KK, Lau SK, Chan KH, Mok KY, Luk HK, Yip CC, Ma YK, Sinn LH, Lam SH, Ngai CW, Hung IF, Chan KH, Yuen KY. 2016. Pulmonary and extrapulmonary complications of human rhinovirus infection in critically ill patients. J Clin Virol 77:85-91.
- 4. Warren-Gash C, Blackburn R, Whitaker H, McMenamin J, Hayward AC. 2018. Laboratory-confirmed respiratory infections as triggers for acute myocardial infarction and stroke: a self-controlled case series analysis of national linked datasets from Scotland. Eur Respir J 51.
- 5. To KK, Lu L, Yip CC, Poon RW, Fung AM, Cheng A, Lui DH, Ho DT, Hung IF, Chan KH, Yuen KY. 2017. Additional molecular testing of saliva specimens improves the detection of respiratory viruses. Emerg Microbes Infect 6:e49.
- 6. To KK, Yip CC, Lai CY, Wong CK, Ho DT, Pang PK, Ng AC, Leung KH, Poon RW, Chan KH, Cheng VC, Hung IF, Yuen KY. 2018. Saliva as a diagnostic specimen for testing respiratory virus by a point-of-care molecular assay: a diagnostic validity study. Clin Microbiol Infect 10.1016/j.cmi.2018.06.009.
- 7. Jain S, Self WH, Wunderink RG, Fakhran S, Balk R, Bramley AM, Reed C, Grijalva CG, Anderson EJ, Courtney DM, Chappell JD, Qi C, Hart EM, Carroll F, Trabue C, Donnelly HK, Williams DJ, Zhu Y, Arnold SR, Ampofo K, Waterer GW, Levine M, Lindstrom S, Winchell JM, Katz JM, Erdman D, Schneider E, Hicks LA, McCullers JA, Pavia AT, Edwards KM, Finelli L, Team CES. 2015. Community-Acquired Pneumonia Requiring Hospitalization among U.S. Adults. N Engl J Med 373:415-427.
- 8. **Kurai D, Saraya T, Ishii H, Takizawa H.** 2013. Virus-induced exacerbations in asthma and COPD. Front Microbiol **4:293**.
- 9. Self WH, Williams DJ, Zhu Y, Ampofo K, Pavia AT, Chappell JD, Hymas WC, Stockmann C, Bramley AM, Schneider E, Erdman D, Finelli L, Jain S, Edwards

- **KM**, **Grijalva CG**. 2016. Respiratory Viral Detection in Children and Adults: Comparing Asymptomatic Controls and Patients With Community-Acquired Pneumonia. J Infect Dis **213**:584-591.
- 10. Kwong JC, Schwartz KL, Campitelli MA, Chung H, Crowcroft NS, Karnauchow T, Katz K, Ko DT, McGeer AJ, McNally D, Richardson DC, Rosella LC, Simor A, Smieja M, Zahariadis G, Gubbay JB. 2018. Acute Myocardial Infarction after Laboratory-Confirmed Influenza Infection. N Engl J Med 378:345-353.
- 11. **Russell E, Yang A, Tardrew S, Ison MG.** 2018. Parainfluenza Virus in Hospitalized Adults: A 7-Year Retrospective Study. Clin Infect Dis 10.1093/cid/ciy451.
- 12. **Blackburn R, Zhao H, Pebody R, Hayward A, Warren-Gash C.** 2018. Laboratory-Confirmed Respiratory Infections as Predictors of Hospital Admission for Myocardial Infarction and Stroke: Time-Series Analysis of English Data for 2004-2015. Clin Infect Dis **67:**8-17.
- 13. Chan PK, Tam WW, Lee TC, Hon KL, Lee N, Chan MC, Mok HY, Wong MC, Leung TF, Lai RW, Yeung AC, Ho WC, Nelson EA, Hui DS. 2015. Hospitalization Incidence, Mortality, and Seasonality of Common Respiratory Viruses Over a Period of 15 Years in a Developed Subtropical City. Medicine (Baltimore) 94:e2024.
- 14. **To KK, Wong SS, Li IW, Hung IF, Tse H, Woo PC, Chan KH, Yuen KY.** 2010. Concurrent comparison of epidemiology, clinical presentation and outcome between adult patients suffering from the pandemic influenza A (H1N1) 2009 virus and the seasonal influenza A virus infection. Postgrad Med J **86:**515-521.
- 15. Hung IF, Zhang AJ, To KK, Chan JF, Zhu SH, Zhang R, Chan TC, Chan KH, Yuen KY. 2017. Unexpectedly Higher Morbidity and Mortality of Hospitalized Elderly Patients Associated with Rhinovirus Compared with Influenza Virus Respiratory Tract Infection. Int J Mol Sci 18.
- 16. **Semret M, Schiller I, Jardin BA, Frenette C, Loo VG, Papenburg J, McNeil SA, Dendukuri N.** 2017. Multiplex Respiratory Virus Testing for Antimicrobial Stewardship: A Prospective Assessment of Antimicrobial Use and Clinical Outcomes Among Hospitalized Adults. J Infect Dis **216**:936-944.
- 17. **World Health Organization.** 2016. WHO Manual for estimating the economic burden of seasonal influenza. Available at http://wwwwhoint/immunization/documents/financing/who\_ivb\_1604/en/ Accessed on 6th October, 2018.
- 18. Miller JM, Binnicker MJ, Campbell S, Carroll KC, Chapin KC, Gilligan PH, Gonzalez MD, Jerris RC, Kehl SC, Patel R, Pritt BS, Richter SS, Robinson-Dunn B, Schwartzman JD, Snyder JW, Telford S, 3rd, Theel ES, Thomson RB, Jr., Weinstein MP, Yao JD. 2018. A Guide to Utilization of the Microbiology Laboratory for Diagnosis of Infectious Diseases: 2018 Update by the Infectious Diseases Society of America and the American Society for Microbiology. Clin Infect Dis 10.1093/cid/ciy381.
- 19. **Kim YG, Yun SG, Kim MY, Park K, Cho CH, Yoon SY, Nam MH, Lee CK, Cho YJ, Lim CS.** 2017. Comparison between Saliva and Nasopharyngeal Swab Specimens for Detection of Respiratory Viruses by Multiplex Reverse Transcription-PCR. J Clin Microbiol **55:**226-233.
- 20. Sbiti-Rohr D, Kutz A, Christ-Crain M, Thomann R, Zimmerli W, Hoess C, Henzen C, Mueller B, Schuetz P, Pro HSG. 2016. The National Early Warning Score (NEWS)

- for outcome prediction in emergency department patients with community-acquired pneumonia: results from a 6-year prospective cohort study. BMJ open **6:**e011021.
- 21. **Centers for Disease Control and Prevention.** Influenza specimen collection desk reference guide. Available at https://www.cdc.gov/flu/pdf/freeresources/healthcare/flu-specimen-collection-guide.pdf. Accessed on 22 February, 2018.
- 22. Benet T, Sanchez Picot V, Messaoudi M, Chou M, Eap T, Wang J, Shen K, Pape JW, Rouzier V, Awasthi S, Pandey N, Bavdekar A, Sanghavi S, Robinson A, Rakoto-Andrianarivelo M, Sylla M, Diallo S, Nymadawa P, Naranbat N, Russomando G, Basualdo W, Komurian-Pradel F, Endtz H, Vanhems P, Paranhos-Baccala G, Global Approach to Biological Research Id, Epidemics in Low-income countries N, Global Approach to Biological Research Id, Epidemics in Low-income countries N. 2017. Microorganisms Associated With Pneumonia in Children <5 Years of Age in Developing and Emerging Countries: The GABRIEL Pneumonia Multicenter, Prospective, Case-Control Study. Clin Infect Dis 65:604-612.